CLINICAL TRIAL: NCT07065474
Title: Effectiveness of Edutainment-Based Interventions in Increasing Knowledge of Rheumatic Fever and Rheumatic Heart Disease Among School-Going Children in Nepal: Study Protocol for Colors to Save Hearts Quasi-Experimental Pretest-Posttest Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu Institute of Child Health (Other)
Responsible Party: Principal Investigator, Shishir Paudel, Monitoring, Evaluation, Accountability, and Learning Officer, Kathmandu Institute of Child Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Color to Save Hearts- KIOCH
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Rheumatic Heart Disease
Keywords: Colour to Save Hearts; Rheumatic heart disease; Rheumatic Fever; Health awarness; Youth intervention
MeSH Terms: conditions — Rheumatic Heart Disease; Rheumatic Fever

STUDY DESIGN:
Intervention Model Description: This study will employ a quasi-experimental pretest-posttest design with a waitlist control group to evaluate the effectiveness of an edutainment-based educational intervention aimed at increasing knowledge about ARF and RHD among school-going children. The design allows for comparisons between the intervention and control groups while ensuring ethical considerations through eventual intervention delivery to all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In the intervention group, students will be exposed to the full package of educational materials (Experimental): Grades 6 to 7 Coloring Book
  With two components:
  * Stories
  * Coloring Assignments • Narratives designed to explain key concepts related to RHD • Activities based on the stories to reinforce learning. Video session • Students will watch educational videos containing information about ARF and RHD, its symptoms, prevention, control, management and treatment.
  Classroom interactive sessions • Discussion and activities designed to engage students and clarify their understanding on ARF and EHD Grades 8 to 9 Activity book
  With two components:
  * Heart Coloring Assignments
  * Games • Heart coloring assignments aims to familiarize participants with the basic structure of human heart • Games includes puzzles, scrambled words, maze run with content on RHD awareness to engaged participants Video session • Students will be exposed to video contain with information regarding ARF and RHD, its symptoms, prevention, control, management and treatment
  Interventions: Other: education material
- Control group (No Intervention): No intervention will be applied

INTERVENTIONS:
Other: education material — For students in Grades 6 to 7, the intervention comprises a coloring book that integrates storytelling and coloring assignments designed to explain key concepts related to ARF and RHD. In addition, students in these grades will watch video sessions that cover the symptoms, causes, prevention, and treatment of ARF and RHD. These videos serve to visualize the information introduced in the books. Complementing these materials, the intervention includes interactive classroom sessions facilitated by the trained field team, during which students will participate in guided discussions and activities to enhance their understanding and retention of health messages. For students in Grades 8 to 9, the intervention uses a more advanced format tailored to older adolescents. These students will receive an activity book that includes heart anatomy coloring assignments and games such as puzzles, scrambled words, and maze runs that incorporate facts and concepts about RHD.
  Arms: In the intervention group, students will be exposed to the full package of educational materials

SUMMARY:
Background: Acute rheumatic fever (ARF) and its sequela, rheumatic heart disease (RHD), remain significant public health concerns in low- and middle-income countries, including Nepal. Despite their preventable nature, awareness of ARF and RHD among schoolchildren is limited. Innovative, age-appropriate health education strategies are urgently needed to promote early recognition and prevention.

Objective: This study aims to evaluate the effectiveness of an edutainment-based intervention in improving knowledge of ARF and RHD among school-going children in Nepal.

Methods: A quasi-experimental pretest-posttest study design with a waitlist control group will be employed across 24 public schools in six diverse districts. A total of 2,400 students from Grades 6 to 9 will be included. The intervention integrates creative educational tools-coloring books, activity books, storytelling, videos, and interactive sessions-tailored to different age groups. Knowledge change will be measured using a validated questionnaire administered at baseline and post-intervention. Secondary outcomes include the prevalence of RHD-related symptoms assessed through clinical screening.

Expected Outcomes: It is hypothesized that students in the intervention group will demonstrate a statistically significant improvement in knowledge scores compared to their baseline levels and the control group. The study will also assess the feasibility and acceptability of the intervention and inform recommendations for broader school-based health education programs.

Conclusion: This study addresses a critical gap in child health education in Nepal using an innovative, scalable approach. Findings will contribute to the evidence base for integrating edutainment into school curricula to combat preventable diseases like RHD in resource-limited settings.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the effectiveness of an edutainment-based educational intervention in improving knowledge about acute rheumatic fever (ARF) and rheumatic heart disease (RHD) among school-going children in Nepal. The secondary aims are to assess the prevalence of RHD-related symptoms among school-going children through basic clinical screening, evaluate the baseline knowledge levels of students regarding ARF and RHD, and measure the effectiveness of the intervention in improving students' knowledge through a quasi-experimental pretest-posttest design.

Based on these aims, the primary hypothesis (H1) is that the edutainment-based intervention will lead to a statistically significant improvement in knowledge scores related to ARF and RHD among schoolchildren in the intervention group when compared to their baseline scores.

Methods Study Design This study will employ a quasi-experimental pretest-posttest design with a waitlist control group to evaluate the effectiveness of an edutainment-based educational intervention aimed at increasing knowledge about ARF and RHD among school-going children.

Study Setting This study will be conducted across six diverse districts of Nepal, selected to represent a range of geographical regions and socio-economic conditions. The chosen districts are Bardiya, Bajhang, Dailekh, Gulmi, Jhapa, and Siraha. Each of these districts includes a mix of urban, semi-urban, and rural areas, allowing the study to capture variation in health awareness, access to education, and healthcare infrastructure. These districts were purposively selected due to their involvement in the PEN-Plus project, an initiative led by the Kathmandu Institute of Child Health (KIOCH). Within each district, one municipality has been selected as the implementation site for the intervention.

Participants selection Inclusion and exclusion criteria This study includes school-going children enrolled in public schools from grades 6 to 9 within the selected municipalities of six districts in Nepal. Students will be eligible for inclusion in the study if they are formally enrolled in one of the selected public schools and are studying in grades 6 to 9 during implementation of this study. To ensure ethical compliance, only those students whose parents or guardians provide written informed consent will be allowed to participate. In addition, assent will be obtained from the students themselves. Students will be excluded from the study if they or their guardians decline to participate or fail to provide the required consent and assent. Students who are absent during both the baseline and post-intervention assessments will also be excluded from the final analysis.

Sample size calculation The sample size was calculated using the formula for comparing paired means, suitable for evaluating changes in knowledge scores before and after an intervention within the same group. The parameters for the calculation included a 95% confidence level (Zα/2 = 1.96), 80% power (Zβ = 0.84). Given the absence of precise prior research findings, and for the purpose of this calculation, the standard deviation of the difference in pre- and post-test scores (σ) was conservatively estimated to be 1. A small to medium effect size (Cohen's d ≈ 0.3) was used for the calculation. Based on these parameters, the minimum required sample size per school was estimated at approximately 87 students. With 12 schools participating in the study (two from each of six districts), the total required sample size across all schools was approximately 1,044 students. Given the cluster sampling design, where students are grouped within schools, this figure was first adjusted for design effect. Assuming an average cluster (school) size of 100 students and an intra-cluster correlation coefficient (ICC) of 0.02, the design effect (DEFF) was calculated as 1 + (100 - 1) × 0.02 = 2.0, increasing the sample size to 2,088 students. Subsequently, a 10% inflation was applied to account for potential non-response, absenteeism, and loss to follow-up, resulting in a final adjusted minimum sample size of 2,400 students. The study will include 12 schools (two from each of the six selected districts, one assigned to the intervention group and one to the waitlist control group). Assuming full enrollment in the selected classrooms, the projected total sample size is approximately 2,469 students, comprising around 1,487 students in the intervention group and 982 in the control group. This slight imbalance in group sizes is due to the constraint that the students within selected classrooms are included, and individual-level randomization is not feasible. Nonetheless, the total projected sample exceeds the adjusted minimum requirement, ensuring adequate statistical power for both primary and subgroup analyses

Sampling procedure A stepwise sampling approach will be employed. In each of the six selected districts, one municipality will be purposively chosen based on the implementation of the PEN-Plus project. In each municipality, two public schools will be selected using a simple random sampling method from the official list of schools. Within each selected school, one classroom from grades 6-7 (lower secondary) and one from grades 8-9 (upper secondary) will be purposively selected in coordination with school authorities based on feasibility and class stability. All students in the selected classrooms will be enrolled through complete enumeration to ensure adequate representation for analysis.

Study Procedure The study will follow a structured implementation process involving orientation, baseline data collection, intervention delivery, midpoint monitoring, endline assessment, and post-intervention delivery to waitlist control schools. These steps will be coordinated by the central research team and executed by trained field researchers, with active collaboration from school staff and medical officers.

Recruitment and Consent Prior to data collection, each selected school will be formally approached for administrative approval. Orientation sessions will then be conducted with school teachers and administrators to familiarize them with the study's objectives, data collection tools, intervention materials, and their expected roles during implementation. Recruitment of participants will occur within selected class sections of Grades 6 to 9 in the participating schools. Prior to enrollment, written informed consent will be obtained from the parents or guardians of all eligible students, and written assent will be obtained from the students themselves. Participation is voluntary, and students may withdraw at any stage without penalty. Only those students who provide both consent and assent will be included in the study.

Randomization and Blinding In each of the six selected municipalities, four public schools will be chosen using a simple random sampling method. Among these, two schools will be assigned to the intervention group, and the other two will serve as the waitlist control group. This school-level allocation ensures feasibility in implementation and minimizes contamination across groups. Although blinding of participants and intervention facilitators is not feasible due to the nature of the intervention, school staff and students will not be informed at the outset about their allocation to either the intervention or control group. This partial concealment is expected to minimize performance and expectation biases during the baseline assessment phase. All data collectors will be trained to apply standardized tools uniformly across both groups, thereby reducing measurement bias.

Intervention In this study, the intervention is stratified by grade level to ensure that the educational content is developmentally appropriate and effectively engages students from different age groups. For students in Grades 6 to 7, the intervention comprises a coloring book that integrates storytelling and coloring assignments designed to explain key concepts related to ARF and RHD. These stories aim to simplify complex health information, while the coloring activities reinforce learning through creative engagement. In addition, students in these grades will watch video sessions that cover the symptoms, causes, prevention, and treatment of ARF and RHD. These videos serve to visualize the information introduced in the books. Complementing these materials, the intervention includes interactive classroom sessions facilitated by the trained field team, during which students will participate in guided discussions and activities to enhance their understanding and retention of health messages. For students in Grades 8 to 9, the intervention uses a more advanced format tailored to older adolescents. These students will receive an activity book that includes heart anatomy coloring assignments and games such as puzzles, scrambled words, and maze runs that incorporate facts and concepts about RHD. The objective of these materials is to stimulate critical thinking and promote deeper engagement with the topic. Like the younger group, students in Grades 8 to 9 will also view educational videos on ARF and RHD and participate in classroom discussions, which will be more analytical and focused on reinforcing prevention messages and encouraging health-seeking behavior

Outcome measurements The primary outcome of the study is the change in knowledge about ARF and RHD among schoolchildren, assessed using a structured questionnaire administered at two time points: baseline (pretest) and end line (posttest). The questionnaire includes items assessing understanding of causes, symptoms, transmission, prevention, and treatment of ARF and RHD. For students in Grades 6 to 8, the tool will be administered via interview to ensure comprehension; students in Grades 9 to 10 will complete a self-administered version of the same instrument. The tool to be used is included structured to cover four major domains: basic knowledge and symptoms, risk factors and prevention, diagnosis and treatment, and impact of the disease. The knowledge scale comprises 14 single-best-answer multiple-choice questions. Each correct response is assigned a score of one, while incorrect and "don't know" responses receive a score of zero. The total knowledge score ranges from 0 to 14, with higher scores indicating better knowledge about ARF and RHD.

To ensure the validity of the instrument, the questionnaire was developed following an extensive review of existing literature on school-based health education and global guidelines related to ARF and RHD. Content validity was established through consultations with subject matter experts in cardiology, community medicine, pediatrics, public health, health education, and school health. Face validity was evaluated by conducting cognitive interviews with a small group of students from Budhanilkantha Municipality to confirm the clarity, appropriateness, and interpretability of the items. Additionally, a pretest was conducted in a public school within the Budhanilkantha Municipality, with approximately 60 students, allowing for refinement of question wording and format based on participant feedback. Internal consistency of the knowledge scale will be examined during the analysis phase using Cronbach's alpha to determine the reliability of the measure.

Statistical Analysis Data will be collected using KoboToolbox and exported to SPSS for statistical analysis. Descriptive statistics will be used to summarize the demographic and baseline characteristics of the participants, including age, sex, academic grade, parental education, district, and the presence of health staff at school. Means and standard deviations will be reported for continuous variables, while frequencies and percentages will be used for categorical variables. To evaluate the primary outcome, changes in knowledge scores before and after the intervention will be assessed using paired t-tests within the intervention group. If the assumption of normality is violated, the Wilcoxon signed-rank test will be used as a non-parametric alternative. Independent t-tests or Mann-Whitney U tests, depending on data distribution, will be used to compare posttest knowledge scores between the intervention and waitlist control groups. For multivariable analysis, posttest knowledge scores will be dichotomized into "high" and "low" categories based on the median score. Binary logistic regression will be employed to examine the association between exposure to the intervention and the likelihood of achieving high knowledge. The regression model will adjust for potential confounding variables, including age, gender, academic grade, parental education, district, family history of RHD, and the presence of a school health nurse. Results will be presented as adjusted odds ratios (AORs) with 95% confidence intervals, and statistical significance will be set at p < 0.05. The internal consistency of the knowledge questionnaire will be assessed using Cronbach's alpha to evaluate the reliability of the scale. Any missing data will be examined, and appropriate imputation techniques will be applied if the proportion of missing responses is substantial.

Program Assessment and Process Evaluation To ensure the reliability and quality of intervention implementation, the study will include a comprehensive assessment of training, supervision, and delivery processes. Prior to data collection and intervention rollout, all field researchers will undergo a standardized training program conducted by the central research team. The training will cover ethical research conduct, consent procedures, administration of data collection tools, delivery of intervention materials, and procedures for midpoint monitoring and reinforcement. Trainers will employ participatory teaching methods such as role-plays, group discussions, and mock classroom sessions to ensure consistent understanding and preparedness among field staff. During the intervention phase, process evaluation will be embedded to monitor the quality, reach, and responsiveness of the educational sessions. Supervisory visits by the central team will be scheduled during the implementation period to observe classroom activities, ensure adherence to standardized delivery protocols, and provide on-site mentoring when needed. Field researchers will maintain structured implementation logs documenting key elements such as the number of sessions completed, duration of each session, material distribution, teacher involvement, and student participation.

In addition to internal monitoring, midpoint visits two weeks after intervention initiation will be used to evaluate student engagement, reinforce key messages, and identify potential barriers to understanding or participation. Feedback from teachers and students will be solicited informally during these visits and documented for process improvement. The consistency of intervention delivery across schools and districts will be assessed through debriefing meetings and progress tracking by the central team, which will ultimately inform recommendations for broader scale-up of the program.

Ethical Considerations This study complies with the national ethical guidelines of Nepal and the international ethical principles outlined in the Declaration of Helsinki. The study has been applied at Institutional Review Board of the Nepal Health Research Council for ethical approval. If any changes are to be made in the study amendment will be made as per the NHRC ethics guideline. Written informed consent will be obtained from the parents or legal guardians of all participating students, and assent will be sought from the students themselves prior to their enrollment in the study. Participants will be informed about the voluntary nature of their participation, their right to withdraw at any point without any consequences, and the measures in place to protect their confidentiality and privacy. All data collected during the study will be anonymized using unique identification codes and stored securely with restricted access, ensuring that no personally identifiable information is disclosed at any stage. Screening for RHD-related symptoms will be respectfully performed by qualified medical officers. Students identified with potential RHD symptoms will be referred for further diagnostic evaluation at designated PEN-Plus clinics. The program will cover necessary transportation and follow-up care costs to eliminate access barriers and ensure ethical equity in health service delivery. To ensure transparency and accountability, regular coordination will be maintained with school authorities, municipal health offices, and parents throughout the study period. Results of the study will be disseminated to stakeholders, including schools, local governments, and health authorities, in a manner that supports informed decision-making and potential scale-up of effective interventions.

ELIGIBILITY:
Inclusion Criteria:

* Students will be eligible for inclusion in the study if they are formally enrolled in one of the selected public schools and are studying in grades 6 to 9 during implementation of this study.

Exclusion Criteria:

* Students will be excluded from the study if they or their guardians decline to participate or fail to provide the required consent and assent. Students who are absent during both the baseline and post-intervention assessments will also be excluded from the final analysis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge about ARF and RHD | 3 months
  The primary outcome of the study is the change in knowledge about ARF and RHD among schoolchildren, assessed using a structured questionnaire administered at two time points: baseline (pretest) and end line (posttest). The knowledge will be assessed by the tool developed by the research team were the knowledge scale comprises 14 single-best-answer multiple-choice questions. Each correct response is assigned a score of one, while incorrect and "don't know" responses receive a score of zero. The total knowledge score ranges from 0 to 14, with higher scores indicating better knowledge about ARF and RHD.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandeepa Karki, MD Community Medicine, Principal Investigator — Kathmandu Institute of Child Health; Mr. Dhurba Khatri, MPH, Principal Investigator — Kathmandu Institute of Child Health; Mr. Shishir Paudel, MPH, Principal Investigator — Kathmandu Institute of Child Health
Locations (1):
- Kathmandu Institute of Child Health, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
To protect the confidentiality of participants informations, individual data will not be share rather grouped data or cleaned data will be shared without the presence of participants identifiers.